CLINICAL TRIAL: NCT05532553
Title: Association Between Carotid Atherosclerosis and Fatty Liver Index in Patients With Type 2 Diabetes Mellitus
Brief Title: Relation Between Carotid Atheroscerosis With DM &Fatty Liver
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ehab Makram, Director, Assiut University
Other Study IDs: Atherosclerosis With DM&fatty
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Atherosclerosis With Diabetes Mellitus and Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patient with T2DM and fatty liver.
  Interventions: Device: Carotid Doppler U/S
- Group 2: patients with fatty liver only ( control group).
  Interventions: Device: Carotid Doppler U/S

INTERVENTIONS:
Device: Carotid Doppler U/S — Measurement of carotid intima media thickness by carotid doppler ultrasound

SUMMARY:
To determine the risk of atherosclerosis in NAFLD patients who have T2DM by meauring Carotid intima media thickness (CIMT) using carotid doppler ultrasound.

DETAILED DESCRIPTION:
Fatty liver is one of the most common chronic liver diseases in the world. It's prevalence is reported to be 10-40% in the adult populations. At least 57% to 80% of them are associated with diabetes (1.2).Atherosclerosis and cardiovascular diseases are also highly prevalent in this group of patients(10).

Non-alcoholic fatty liver disease ( NAFLD) is characterized pathophysiological by hepatic fat accumulation independent of excessive alcohol use(3.4). Fatty liver index (FLI) has been demonstrated good diagnostic accuracy in different populations(6.7)...FLI will be based on BMI, waist circumference (WC), triacylglycerols (TG) and g-glutamyl transferase (GGT).

The individuals with NAFLD have a higher risk of 10-year cardiovascular events than healthy individuals.(10) .NAFLD and T2DM are common conditions that regularly co-exist and can act synergistically to drive adverse outcomes(5). Diabetic macrovascular complications are the major chronic complications and the leading cause of death among the patients with T2DM, of which the pathological basis is atherosclerosis.(8) Atherosclerosis usually starts in the vascular intima, progressing to the medial arterial wall(9).Carotid intima-media thickness (CIMT) is an indicator of the risk of vascular disease. Increased CIMT and presence of atherosclerotic plaque are considered as a reliable ultrasound biomarker of subclinical atherosclerosis and can be used for cardiovascular risk assessment[9].

In this study the investigators have the aim of evaluating the possible association between non-invasive index of fatty liver (FLI) and the presence of carotid atherosclerosis in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fatty liver (diabetic& not diabetic).

Exclusion Criteria:

* 1-Other causes of Liver disease ( (viral hepatitis, drug-induced liver disease, hepatolenticular degeneration, autoimmune liver disease, schistosomiasis liver disease, cirrhosis, etc.) 2- Heavy smoker.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who will be presented to internal medicine department& outpatient clinics at Assiut university hospital divided into 2 groups.
  Group 1:Patient with T2DM and fatty liver. Group 2: patients with fatty liver only ( control group). Carotid doppler ultrasonography will be considered for both groups to measure Carotid Intima Media Thickness (CIMT).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of carotid atherosclerosis | baseline
  To determine the risk of atherosclerosis in NAFLD patients who have T2DM by measuring CIMT using carotid doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Anwar Mohamed Khalifa, Doctor, Study Director — Assiut University

REFERENCES:
- [Background] Pereira K, Salsamendi J, Casillas J. The Global Nonalcoholic Fatty Liver Disease Epidemic: What a Radiologist Needs to Know. J Clin Imaging Sci. 2015 May 29;5:32. doi: 10.4103/2156-7514.157860. eCollection 2015. PMID 26167390
- [Background] Younossi ZM. Non-alcoholic fatty liver disease - A global public health perspective. J Hepatol. 2019 Mar;70(3):531-544. doi: 10.1016/j.jhep.2018.10.033. Epub 2018 Nov 9. PMID 30414863
- [Background] Benedict M, Zhang X. Non-alcoholic fatty liver disease: An expanded review. World J Hepatol. 2017 Jun 8;9(16):715-732. doi: 10.4254/wjh.v9.i16.715. PMID 28652891
- [Background] Rinella ME, Sanyal AJ. NAFLD in 2014: Genetics, diagnostics and therapeutic advances in NAFLD. Nat Rev Gastroenterol Hepatol. 2015 Feb;12(2):65-6. doi: 10.1038/nrgastro.2014.232. Epub 2015 Jan 6. PMID 25560844
- [Background] Hazlehurst JM, Woods C, Marjot T, Cobbold JF, Tomlinson JW. Non-alcoholic fatty liver disease and diabetes. Metabolism. 2016 Aug;65(8):1096-108. doi: 10.1016/j.metabol.2016.01.001. Epub 2016 Jan 11. PMID 26856933
- [Background] Lee JH, Kim D, Kim HJ, Lee CH, Yang JI, Kim W, Kim YJ, Yoon JH, Cho SH, Sung MW, Lee HS. Hepatic steatosis index: a simple screening tool reflecting nonalcoholic fatty liver disease. Dig Liver Dis. 2010 Jul;42(7):503-8. doi: 10.1016/j.dld.2009.08.002. Epub 2009 Sep 18. PMID 19766548
- [Background] Bedogni G, Bellentani S, Miglioli L, Masutti F, Passalacqua M, Castiglione A, Tiribelli C. The Fatty Liver Index: a simple and accurate predictor of hepatic steatosis in the general population. BMC Gastroenterol. 2006 Nov 2;6:33. doi: 10.1186/1471-230X-6-33. PMID 17081293
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Stein JH, Tattersall MC. Carotid intima-media thickness and cardiovascular disease risk prediction. J Am Coll Cardiol. 2014 Jun 3;63(21):2301-2. doi: 10.1016/j.jacc.2014.02.528. Epub 2014 Mar 5. No abstract available. PMID 24613323
- [Background] Wojcik-Cichy K, Koslinska-Berkan E, Piekarska A. The influence of NAFLD on the risk of atherosclerosis and cardiovascular diseases. Clin Exp Hepatol. 2018 Mar;4(1):1-6. doi: 10.5114/ceh.2018.73155. Epub 2018 Jan 20. PMID 29594192